CLINICAL TRIAL: NCT00074464
Title: Cholesterol Homeostasis in Framingham Offspring Study
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1242; R01HL074388 (NIH)
Record Dates: First submitted 2003-12-12; First posted 2003-12-15 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Atherosclerosis; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Atherosclerosis; Coronary Disease

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
To investigate the predictive value of using measures of cholesterol homeostasis to identify individuals at high risk of developing cardiovascular disease relative to established risk factors.

DETAILED DESCRIPTION:
BACKGROUND:

Cholesterol is a major risk factor for coronary heart disease. The current approach to assessing this risk factor is to measure levels in the blood as if blood levels were a static and fixed phenomenon. Cholesterol levels in the blood are in fact a complex product of transport of cholesterol and lipids into and out of various compartments: (1) from the gut, liver or periphery into the blood; (2) from the blood into the periphery and the liver; (3) de novo synthesis of cholesterol in the liver; and (4) excretion from the liver as bile acids. It is possible that one or more of these processes may serve as better risk factors for atherosclerosis or coronary events than simple measures of cholesterol. This study addresses a new and potentially important question.

The study will utilize plasma samples from subjects participating in Cycle 6 of the Framingham Offspring Study. The Framingham Offspring Study is a longitudinal community based study initiated in 1971. A sample of 5,135 men and women, consisting of the offspring of the original Framingham Heart Study and their spouses were enrolled for the study, the objective of which was to identify common factors or characteristics that contribute to cardiovascular disease (CVD) by following its incidence over a long period of time in a large group of participants who had not yet developed overt symptoms of CVD or suffered a heart attack or stroke.

DESIGN NARRATIVE:

The project includes a case-control study relating the new lipid findings to cardiovascular disease (CVD), a cross-sectional study to establish normal values and associations with diet and genotypes, and a prospective study of cardiovascular events during a 10-year follow-up period. The specific aims are to 1) quantify circulating indicators of cholesterol homeostasis [levels of phytosterols and cholestanol (surrogate measures of cholesterol absorption) and cholesterol precursors (surrogate measures of cholesterol synthetic rates)] in plasma samples from Framingham Offspring Study participants diagnosed with established CVD and/or >50% carotid stenosis (N=165) not taking lipid-lowering medication and control subjects matched for age, sex, body mass index, hypertension and smoking status (n=330); 2) evaluate the validity of using indicators of cholesterol homeostasis to predict CVD risk in the Framingham Offspring Study-Cycle 6 participants by a) establishing adult normal ranges for circulating levels of phytosterol, cholestanol and cholesterol precursor (N=3378), b) defining the relationship between phytosterol, cholestanol and cholesterol precursor levels, and lipid, lipoprotein and apolipoprotein levels in plasma, c) defining the relationship between phytosterol, cholestanol and cholesterol precursor levels and selected dietary intake data (energy, protein, fat, saturated, monounsaturated, polyunsaturated and trans fatty acids, cholesterol, fiber and antioxidant supplements) and d) determining the relationship between phytosterol, cholestanol and cholesterol precursor levels and selected genotype data related to CVD risk (gene loci of apo E, apo A-IV, scavenger receptor class B type 1 [SRB1], and ATP-binding cassette [ABC] G5 and ABCG8 transporters); and 3) monitor clinical events in the Framingham Offspring Study cohort throughout a 10-year period (1995-2005) and relate these data to the phytosterol, cholestanol and cholesterol precursor levels. Measures of cholesterol homeostasis will be quantified first in subjects identified in specific aim #1 and then the balance of subjects identified in specific aim #2, achievable now due to the development of a gas chromatographic method using a single plasma sample. These data will be assessed relative to dietary, biochemical and genotype data currently available for the cohort. The results of the study will define the relationship between markers of cholesterol absorption and synthesis, and CVD outcomes; establish reference values for measures of cholesterol absorption and synthesis; and assess the predictive value of these measures to identify high risk individuals relative to established risk factors.

ELIGIBILITY:
No eligibility criteria

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Framingham Offspring Study Cycle 6 Participants
Sampling Method: Probability Sample
Enrollment: 3378 (Actual)
Dates: Start 2003-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
quantification of circulating indicators of cholesterol homeostasis | 1 time point
  phytosterols and cholestanol (surrogate measures of cholesterol absorption) cholesterol precursors (surrogate measures of cholesterol synthetic rates)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Lichtenstein, Principal Investigator — Tufts University

REFERENCES:
- [Derived] Matthan NR, Zhu L, Pencina M, D'Agostino RB, Schaefer EJ, Lichtenstein AH. Sex-specific differences in the predictive value of cholesterol homeostasis markers and 10-year cardiovascular disease event rate in Framingham Offspring Study participants. J Am Heart Assoc. 2013 Feb 19;2(1):e005066. doi: 10.1161/JAHA.112.005066. PMID 23525441